CLINICAL TRIAL: NCT00136617
Title: Comparison of a Fixed-Schedule Therapy Versus a Symptom-Triggered Therapy for Alcohol Withdrawal Syndrome in Medical Out-Patients
Brief Title: Outpatient Treatment of Alcohol Withdrawal Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AWS
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2009-03-02 (Estimated); Status verified 2009-02

CONDITIONS: Alcoholism; Alcohol Withdrawal
Keywords: Short Alcohol Withdrawal Scale; Documentation
MeSH Terms: conditions — Alcoholism | interventions — Chlordiazepoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: chlordiazepoxide

SUMMARY:
The purpose of this study is to compare a fixed-schedule therapy versus a symptom-triggered therapy for alcohol withdrawal syndrome in medical outpatients.

Objectives:

* Self-governance in monitoring AWS (alcohol withdrawal syndrome) symptoms and medication
* Clinically controlled trial of two regimens for medical treatment of alcohol withdrawal syndrome
* Outpatient treatment of alcohol withdrawal syndrome

DETAILED DESCRIPTION:
The objective of this study is to compare a fixed-schedule therapy versus a symptom-triggered therapy for alcohol withdrawal syndrome in medical outpatients.

Objectives:

* Self-governance in monitoring AWS (alcohol withdrawal syndrome) symptoms and medication
* Clinically controlled trial of two regimens for medical treatment of alcohol withdrawal syndrome
* Outpatient treatment of alcohol withdrawal syndrome

Patients and Methods:

This study is a prospective analysis of patients admitted to a medical outpatient clinic between August 25, 2003 and July 1, 2006, who experienced AWS. This study is conducted at Copenhagen Hospital Corporation in Copenhagen, Denmark. Patients were divided into two randomized groups: a symptom-triggered treatment versus a fixed-schedule treatment (known) with chlordiazepoxide. They were diagnosed with AWS according to DSM-IV (Diagnostic and Statistical Manual of Mental Disorders Fourth Edition). They were diagnosed with alcohol dependence according to the ICD-10 (International Statistical Classification of Diseases and Health Related Problems).

Methods:

One hundred fifty consecutive patients who fulfill the inclusion criteria and not the exclusion criteria were offered to participate in the study, i.e. also patients who were detoxified at home or during admission. Patients were scored according to the DSM-IV for AWS and ICD-10 for alcohol dependence, and then they filled out a SAWS (Short Alcohol Withdrawal Scale). The score of 12 was the significant number of splitting patients to mild or moderate AWS. Randomization was done by the Research Unit. Patients were then treated with the traditionally fixed-schedule therapy (day 1, 200mg, chlordiazepoxide decreasing with 25 mg a day) or the new symptom-triggered therapy (up to 300 mg, chlordiazepoxide a day). For up until 10 days, patients monitored themselves for all ten days according to the SAWS. They were asked about mental conditions day 1-14 and every third month using the World Health Organization (WHO)-5 schedule.

On day 10 they filled out an adverse reactions questionnaire on chlordiazepoxide and a DTSQ (Diabetes Treatment Satisfaction Questionnaire) and an ASI (Addiction Severity Index) every third month.

Relapses and intake of any alcohol during a year are monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 18
* Fulfilled informed consent
* Abstained from alcohol within the last 72 hours.
* Agree on both treatment regimens.
* Abstinence during 10 days (monitoring and medication period), i.e. treatment with disulfiram or oral alcometer test on every attendance (Lion Alcometer S-D2).

Exclusion Criteria:

* Oral alcoholmeter test > 0.1.
* Treatment of AWS within the last week
* 3 earlier attempts at outpatient detoxification within the last 2 months without success.
* Allergy or adverse reactions to chlordiazepoxide
* Treatment with medication in interaction with chlordiazepoxide
* Psychiatric comorbidity within the last year, dependence on other drugs except nicotine dependence
* Medically severe comorbidity, especially severe liver insufficiency
* Severe cardiovascular diseases, NIDDM and IDDM.
* A history within the last year of seizures and delirium tremens.
* Patients should be cooperative in terms of cooperation and understanding of the Danish language.
* Females of fertile age without safe contraception, (i.e. IUD, hormone tablets or sterilisation) also pregnant or breastfeeding women were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2003-08; Primary Completion 2006-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To shorten the AWS-period by determining the time to Short Alcohol Withdrawal Scale (SAWS)-score is below 12
To give the most safe treatment to the patients and reduce the risk of further development of alcohol withdrawal syndrome with seizures and delirium tremens
AWS score day 1, 2, 3, etc.
Use of medication
Patient satisfaction
Wellbeing

SECONDARY OUTCOMES:
Compliance in alcohol treatment
Time to first relapse

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Becker, MD, Study Director — Hvidovre University Hospital
Locations (1):
- Alcohol Clinics at Hvidovre Hospital, Hvidovre, Denmark